CLINICAL TRIAL: NCT03583762
Title: Comparison of Time to Appropriate Antibiotic Between Using Microarray Assay and Mass Spectrometry Technique for Identification of Positive Blood Cultures
Brief Title: Time to Appropriate Antibiotic Between Using Microarray Assay and Mass Spectrometry Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Romanee Chaiwarith, Associate Professor, Chiang Mai University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MED-2561-05383
Record Dates: First submitted 2018-06-15; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Septicemia
Keywords: Microarray Assay Technique; Mass Spectrometry Technique; Time to appropriate antibiotic
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention group (Experimental): 100 participants received empiric antibiotic by ID physician, bacterial identification by Mass spectrometry technique
  Interventions: Diagnostic Test: Mass spectrometry
- Post-intervention group (Experimental): 100 participants received empiric antibiotic therapy by ID physician, bacterial identification by Microarray assay from blood culture and confirm with Mass spectrometry technique
  Interventions: Diagnostic Test: Microarray assay

INTERVENTIONS:
Diagnostic Test: Mass spectrometry — Molecular diagnostic test for bacterial identification from bacterial colony
  Arms: Pre-intervention group
Diagnostic Test: Microarray assay — Bacterial identification by Microarray assay from positive blood culture and confirmed by Mass spectrometry technique from bacterial colony. Adjusted antibiotic therapy according to AST Re-evaluation after treatment
  Arms: Post-intervention group

SUMMARY:
This is an experimental study of participants who had positive blood culture to compare time to appropriate antibiotic between using Microarray Assay and Mass Spectrometry to bacterial Identification.

DETAILED DESCRIPTION:
Between June to Dec 2018, 200 participants those met the eligibility criteria were enrolled in this study that is a quasi experimental study. All participants were empirical antibiotic therapy by infectious physician. 100 patients in Pre-intervention group had bacterial identification by Mass spectrometry technique from bacterial colony and 100 patients in Post-intervention group had bacterial identification by Microarray assay from blood culture. Antibiotic adjustment were considered after bacterial identification and result of antibiotic susceptibility testing. Then all participants were re-evaluated outcome after treatment. Finally, the results were ready to analysis in January 2019.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year old with positive hemoculture between June 2018 and Dec 2018
* Internal medicine wards patients at Maharaj Nakorn Chiang Mai Hospital
* Ability to provide informed consent

Exclusion Criteria:

* Suspected contaminated positive blood culture
* Bacteremia cause by more than two species of bacteria, as suspected from the gram staining examinations
* Terminally ill patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07-30 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
To compare the time to appropriate antibiotic therapy in patients with positive blood cultures between using Microarray assays versus Mass Spectrometry technique for Identification of Positive Blood Cultures | 4 days from positive hemoculture
  Comparison of time that participants received appropriate antibiotic therapy between 2 study period (Mass spectrometry technique and Microarray assay group)

SECONDARY OUTCOMES:
Mortality rate at 2 weeks | 14 days from positive hemoculture
  To compare proportion of mortality between 2 study periods (Mass spectrometry technique and Microarray assay group) at 2 weeks after enrollment
Length of hospital stays | 30 days
  To compare lengths of hospital stay between 2 study periods (Mass spectrometry technique and Microarray assay group)
Cost of antibiotic therapy | 14 days
  To compare the cost of antibiotics for the course of treatment during study period between 2 study period (Mass spectrometry technique and Microarray assay group)
Percentage of De-escalation or escalation antibiotic | 14 days
  To compare percentage of De-escalation or escalation antibiotic between 2 study periods (Mass spectrometry technique and Microarray assay group)

CONTACTS AND LOCATIONS:
Overall Officials: Parichart Sakulkonkij, MD, Principal Investigator — Chiang Mai University
Locations (1):
- Maharaj Nakorn Chiang Mai Hospital, Department of Medicine, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided